CLINICAL TRIAL: NCT04545840
Title: Prospective Study of Neodent® Implantable Devices of Zirconia System
Brief Title: Prospective Neodent® Zirconia System Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Neodent (Industry)
Responsible Party: Sponsor
Other Study IDs: CS.O.010
Record Dates: First submitted 2020-09-04; First posted 2020-09-11 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Jaw, Edentulous; Jaw, Edentulous, Partially
Keywords: Dental Implants; Mouth Rehabilitation
MeSH Terms: conditions — Jaw, Edentulous; Jaw, Edentulous, Partially | interventions — Dental Implants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- Study group: Zirconia Implants will be placed. More than one implant can be placed in the same patient, as long as the subject presents natural teeth adjacent to the implant site.
  Interventions: Device: Dental Implants

INTERVENTIONS:
Device: Dental Implants — Dental Implants will be used according to standard routine in daily practice, according to all indications as specified by the manufacturer in the IFU (informations for use).

SUMMARY:
The Neodent® Zirconia Implant is designed for the treatment of oral endosteal implantation for the functional and aesthetic rehabilitation, allowing for treatment of patients with different bone qualities.

The objective of the study is to assess the success and survival rates of implantable devices of the Zirconia System, in order to confirm the long-term safety and clinical performance of implants and abutments of the Zirconia System in daily dental practice setting.

Devices will be used according to standard routine in daily practice, according to manufacturer indications in the IFU. Patients will be followed for 36 months after implant placement.

DETAILED DESCRIPTION:
The study protocol was reviewed and approved by an Ethics Committee (CE) in Brazil. The sample will be prospectively and consecutively selected and will consist of patients who are 18 years of age or older, who are in need of and who qualify for single dental implants placement in the posterior maxilla region with Neodent® Zirconia. Informed consent in writing will be obtained from each patient participating in the study prior to any study related procedure.

As this study will be analyzed descriptively, sample size calculation was not performed. To generate reliable results, a total number of 30 implants was assumed to be sufficient. Estimating a rate of 1 implant per patient and a drop-out rate of 15%, a sample size of 36 patients resulting in an estimated number of 36 implants is thought to be sufficient to allow for a descriptive analysis of clinical outcome data up to 36 months after implant placement.

Treatment provided to the subjects will be the responsibility of an appropriately qualified dental practitioner to provide the relevant patient care under clinical study conditions. Zirconia Implants will be placed under local anesthesia and with adequate bone bed preparation in posterior maxilla region. More than one implant can be placed in the same patient, as long as the subject presents natural teeth adjacent to the implant site.

Immediately after implant placement, the final placement torque will be registered. The immediate loading will be applied within 48 hours with the insertion of a provisional prosthesis made from intraoral scanning or scanning of dental casts obtained by conventional impression. The insertion torque shall reach at least 35 N.cm and the subject must have physiologic occlusion to immediate loading. If the patient does not reach the minimum torque (35 N.cm), the patient will be followed until the study end but will not be considered to final statistic or, a different implant line would be placed and the study termination form will be filled. The principal investigator will choose how to procedure in this situation. The selection of the prosthetic component shall be conducted according to the need of each subject and to the manufacturer's instructions (IFU). The final prosthesis will be placed 2 months after implant loading.

Data concerning the studied variables will be collected following the procedures and assessments plan by fulfilling the Case Report Form (CRF), in the following stages: screening (First visit); TP - Implant(s) placement and impression/scanning for temporary prosthesis preparation; T0 - Implant(s) loading (up to 48h after placement); TF - Final prosthesis placement (2 months ± 1 week after loading); T6, T12, T24, T36 - 6, 12, 24 e 36 ± 1 month, respectively, after loading.

Standardized digital periapical radiographs will be obtained in a usual daily practice frequency, as determined by the investigator: at pre-operative, to assess the ridge height and width of the supporting bone and locate major anatomical features; in post-surgery (TP) and in T0, TF, T6, T12, T24 and T36 to verify prosthesis adaptation and osseointegration. Computed tomography scans will be obtained from the region of interest prior to surgery, for the selection of the implant to be inserted.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* Maxillary posterior teeth missing, with adjacent natural teeth;
* Patient who are in need of oral rehabilitation with dental implants and single prostheses and qualify for placement of Zirconia Implants.

Exclusion Criteria:

Subjects under 18 years of age, pregnant or breastfeeding women. And patients that present the device contraindications according to the IFU (instructions for use):

* Signs of allergy or hypersensitivity to the chemical ingredients of the material: Zirconia (Y-ZTP), Zirconium dioxide (ZrO2), Yttrium oxide (Y2O3), Hafnium dioxide (HfO2), Aluminum oxide (Al2O3);
* Acute inflammatory or infectious processes;
* Unsuitable bone volume or quality;
* Serious medical problems (e.g. bone metabolism disorders, blood clotting disorders, unsuitable healing capacity);
* Incomplete jawbone growth;
* Patient uncooperative and not motivated;
* Hypochondria;
* Alcoholism;
* Psychosis;
* Prolonged functional disorders which resist any treatment with medications;
* Xerostomia;
* Weakened immunological system;
* Diseases which require regular use of steroids;
* Uncontrolled endocrine diseases;
* Insufficient oral hygiene;
* Pregnancy;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients 18 years of age or older who are in need of and who qualify for single dental implants placement in the posterior maxilla region with Neodent® Zirconia Implants.
  Patients that give written informed consent to participate in this clinical study.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2020-09-10 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Implant survival rate | 36 months after implant placement
  Implant survival will be defined as no loss of the implant.
Implant success rate | 36 months after implant placement
  Evaluation of implant success will be assessed based on the criteria proposed by Buser et al. (1990).

SECONDARY OUTCOMES:
Implant survival rate | 6 months after implant placement
  Implant survival will be defined as no loss of the implant.
Implant success rate | 6 months after implant placement
  Evaluation of implant success will be assessed based on the criteria proposed by Buser et al. (1990).
Prosthetic survival rate | 36 months after implant placement
  Prosthetic survival will be assessed as the final prosthesis remaining in situ, irrespective of its condition.
Prosthetic success rate | 36 months after implant placement
  Success will be defined as the prosthesis that remained unchanged and did not require any intervention, except routine occlusal adjustments, during the entire observational period
Patient satisfaction: questionnaire | At screening visit, after the temporary prosthesis period and 6, 12, 24 and 36 months after implant placement
  OHIP-14 questionnaire will be used to assess Oral Health Related Quality of Life (OHRQoL), as a measure of patient satisfaction with treatment. Patients will be asked how frequently they have been experiencing the problems assessed by the questionnaire. Small values mean a better quality of life.
Clinician satisfaction: questionnaire | At implant placement, implant loading and 6, 12, 24 and 36 months after implant placement
  The assessment will be performed by means of a questionnaire using a visual analog scale (VAS) in the form of a 10 cm horizontal line, where 0 (left end) indicates minimum satisfaction and 10 (right end) indicates maximum satisfaction. The clinician will be instructed to mark the position considered to best represent their degree of general satisfaction with patient treatment. The score will be measured in centimeters from the left end of the line to the marked point.
Rate of adverse events related to the implant, prosthesis, surgery and oral health | At implant placement, implant loading, final prosthesis placement and 6, 12, 24 and 36 months after implant placement
  Determined by inquiring with the patient and clinical evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Larissa Trojan, PhD, Study Chair — Neodent
Locations (1):
- Instituto Latino Americano de Pesquisa e Ensino Odontológico (ILAPEO), Curitiba, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No